CLINICAL TRIAL: NCT02696083
Title: A Multicenter, Open-Label, Single-Arm, Proof of Concept Study of Pulsed Electromagnetic Field (PEMF) Therapy to Evaluate Synovial Fluid Markers in Subjects With Osteoarthritis of the Knee
Brief Title: Proof of Concept Study of PEMF (Pulsed Electromagnetic Field) Therapy in Subjects With Osteoarthritis of the Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regenesis Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RBI.2015.004
Record Dates: First submitted 2016-02-17; First posted 2016-03-02 (Estimated); Results first posted 2018-01-12 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2017-12

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active Treatment (Experimental)
  Interventions: Device: Provant Therapy System

INTERVENTIONS:
Device: Provant Therapy System

SUMMARY:
To investigate the effect of PEMF treatment when administered twice daily over a 90-day period by looking at synovial fluid in subjects with osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria:

1. Subject age is greater than or equal to 45 years and less than 80 years of age.
2. Subject has documented Kellgren-Lawrence radiograph score of 2, 3, or 4. Attempts will be made to include at least 3 subjects in each category.
3. Subject is on a stable analgesic regimen for at least two weeks prior to the Screening Visit and anticipates being able to remain on that regimen throughout the study.
4. Subject is willing and able to give written informed consent and to comply with all parts of the study protocol.
5. Female subjects must be post-menopausal, surgically sterile, abstinent, or practicing (or agree to practice) an effective method of birth control if they are sexually active for the duration of the study. (Effective methods of birth control include prescription hormonal contraceptives, intrauterine devices, double-barrier methods, and/or male partner sterilization).

Exclusion Criteria:

1. Subject has documented Kellgren-Lawrence radiograph score of 1.
2. Subject has undergone viscosupplementation treatment for the knee within 2 months of the Screening Visit.
3. Subject has had a total or partial knee replacement.
4. Subject has used topical or oral steroids within 2 months of the Screening Visit.
5. Subject has undergone any anesthetic injection into the knee within 30 days prior to the Screening Visit or within 6 weeks prior to the Screening Visit for long acting lidocaine injection products.
6. Subject has other diseases of the knee joint including inflammatory arthritis (i.e., rheumatoid arthritis, spondyloarthritis, gout and pseudogout), autoimmune disease (i.e., connective tissue disorders), septic arthritis, previous knee injury or intra-articular fracture.
7. Subject will be unable to treat daily over the course of the 90 day treatment period (e.g., travelling without the ability to take Provant).
8. Subject has received any investigational drug or device within 30 days or 5 half-lives of the drug, whichever is longer, prior to the Screening Visit or is enrolled in another clinical trial.
9. Subject has a history of a solid tumor that is not in complete remission for greater than 2 years other than successfully treated non-metastatic basal cell or squamous cell carcinomas of the skin in the treatment area.
10. Subject has a history of blood cancer (e.g., leukemia, lymphoma, multiple myeloma).
11. Subject has an ongoing painful condition, other than osteoarthritis, that in the opinion of the investigator might have a confounding influence on the safety or effectiveness analyses for this study.
12. Subject has a Body Mass Index (BMI) > 38 kg/m2.
13. Subject has a serious psychosocial co-morbidity.
14. Subject has a history of drug or alcohol abuse within one year prior to screening.
15. Subject has an implanted pacemaker, defibrillator, neurostimulator, spinal cord stimulator, bone stimulator, cochlear implant, or other implanted device with an implanted metal lead(s).
16. Subject is currently pregnant or planning on becoming pregnant prior to Day 90.
17. Subject is unwilling or unable to follow study instructions, or comply with the treatment regimen, study visits, and diary entries.
18. Subject is in current litigation regarding knee pain or is receiving Worker's Compensation.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-02-02 (Actual); Primary Completion 2016-09-23 (Actual); Study Completion 2016-09-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Colorado Orthopaedics, Lone Tree, Colorado
  - Spokane Joint Replacement, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Treatment (Provant Therapy System): Provant Therapy System
Period: Overall Study
Arm/Group | Active Treatment (Provant Therapy System)
Started | 19
Completed | 13
Not Completed | 6

BASELINE CHARACTERISTICS:
Groups:
- Active Treatment: Provant Therapy System
Arm/Group | Active Treatment
Number analyzed (Participants) | 19
Age, Continuous [Mean (Full Range); unit: years] | 63.68 [46 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Synovial Markers Showing a Reduction From Baseline Following Treatment at Days 45 and 90
Description: Synovial markers measured included bone morphologic proteins, related proteins Activin A, Osteoactivin, sonic hedgehog, Dickkopf, interleukin cytokines and tumor necrosis factor alpha, Growth Factors and Related Proteins fibroblast growth factors 1,2, androgen receptor, platelet derived growth factor BB, tumor growth factor beta, osteprogenerin, osteopontin, and Insulin like growth factor-1. Inflammation related proteins assayed were monocyte chemoattractant protein-1, macrophage colony-stimulating factor, macrophage inflammatory protein, receptor activator of Nuclear factor κ, and TNF related activation induced cytokine. Adhesion and matrix metalloproteinase proteins levels were also determined. The mean protein concentration was calculated for these markers at Baseline (n=19), Day 45 (n=7) and Day 90 (n=6).
Time Frame: Baseline, Days 45 and 90
Population: The mean protein concentration was calculated for these markers at Baseline (n=19), Day 45 (n=7) and Day 90 (n=6).
Measure: Count of Units; unit: protein markers
Units Other Than Participants: protein markers
Groups:
- BMP and Related Proteins: BMP and related protein synovial markers measured included 9 markers: bone morphologic proteins (BMP-2, BMP-4, BMP-6, BMP-7, BMP-9) and related proteins Activin A, Osteoactivin (Ostact), sonic hedgehog (Shh N) and Dickkopf (DKK-1).
- Cytokines: The 7 synovial markers measured included the levels of interleukin cytokines and tumor necrosis factor alpha (Il-1α, IL-1β, IL-6, IL-8, IL-11, IL-17 and TNFα),
- Growth Factors and Related Proteins: The 10 synovial markers included in this group include Growth Factors and Related Proteins fibroblast growth factors 1,2, androgen receptor, platelet derived growth factor BB, tumor growth factor beta, osteprogenerin, osteopontin, and Insulin like growth factor-1 (FGF-1, FGF-2, AR, PDGF BB, TGF b1, TGF b2, TGF b3, OPG, OPN and IGF-1
- Bone Remodeling Related Proteins: The 6 synovial fluid markers in this group included monocyte chemoattractant protein-1, macrophage colony-stimulating factor, macrophage inflammatory protein, receptor activator of Nuclear factor κ, and TNF related activation induced cytokine (MCP-1, M-CSF, MIP-1a, RANK, TRANCE).
- Adhesion and Matrix Proteins: This group includes 4 adhesion and matrix metalloproteinase proteins: ICAM-1, P-CadH, VCAM-1, and VE-CadH.
- MPP Proteins: The 4 matrix metalloproteinase proteins analyzed in this group include the following: MMP-2, MMP-3, MMP-9, and MMP-13.
Arm/Group | BMP and Related Proteins | Cytokines | Growth Factors and Related Proteins | Bone Remodeling Related Proteins | Adhesion and Matrix Proteins | MPP Proteins
Number analyzed (Participants) | 19 | 19 | 19 | 19 | 19 | 19
Number analyzed (protein markers) | 9 | 7 | 10 | 6 | 4 | 4
protein markers
  Day 45 -# of markers that decreased from Baseline: number analyzed (Participants) | 7 | 7 | 7 | 7 | 7 | 19
  Day 45 -# of markers that decreased from Baseline | 6 | 6 | 8 | 5 | 3 | 2
  Day 90 - # of markers that decreased from Baseline: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
  Day 90 - # of markers that decreased from Baseline | 8 | 7 | 10 | 4 | 4 | 4

ADVERSE EVENTS:
Arm/Group | Active Treatment
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 10/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Treatment (N=19)
Increased knee pain (Musculoskeletal and connective tissue disorders) | 9 (10)
Increase knee swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Exacerbation of patients end stage renal failure (Renal and urinary disorders) | 1 (1)
Anterior C6-C7 Cervical Diskectomy and Fusion with Partial Laminectomy, Medial facetectomy and foram (Musculoskeletal and connective tissue disorders) | 1 (1)
Left knee buckled (Musculoskeletal and connective tissue disorders) | 1 (1)
Prominent Menieres Episode (Ear and labyrinth disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication Rights. Independent analysis and/or publication of data generated or arising from the performance of this Agreement is not permitted without the prior written consent of Regenesis. Such consent may be contingent on Regenesis' review and approval of any proposed analysis and manuscript. Institution will retain the right to review and analyze the database created from this study for its own scientific purposes so long as such scientific purposes are non-commercial in nature.